CLINICAL TRIAL: NCT07252635
Title: Comparison of the DNS-Based Developmental Exercise and Single Leg Squat Exercise on Quadriceps Muscle Activation in Fencers
Brief Title: Comparison of DNS-Based Developmental Exercise and Single Leg Squat Exercise in Fencers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Seda Uluşahin, Assistant Professor, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-1206
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Quadriceps Muscle
Keywords: Exercise; One leg squat; DNS; EMG; Muscle activation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fencers Performing Three Exercises (Experimental): All participants are competitive fencers who will perform three different lower-extremity exercises during the study session. The exercises are:
  Single-leg decline squat
  Single-leg decline squat with core activation
  Half high kneeling exercise based on Dynamic Neuromuscular Stabilization (DNS)
  Each exercise is performed on the dominant leg, following standardized timing in three phases (eccentric, isometric, concentric). The order of exercises is randomized. Muscle activity of the quadriceps (vastus medialis obliquus, vastus lateralis, and rectus femoris) is recorded with surface electromyography (EMG) during all exercises.
  Interventions: Other: EMG analysis during Single-Leg Decline Squat

INTERVENTIONS:
Other: EMG analysis during Single-Leg Decline Squat — EMG analysis during Half high kneeling exercise

SUMMARY:
The goal of this clinical trial is to learn how three different exercises affect quadriceps muscle activity (Vastus medialis, Vastus lateralis, and Rectus femoris) in young fencers. The three exercises are: a single-leg decline squat, a single-leg decline squat with core activation, and a half high-kneeling exercise based on Dynamic Neuromuscular Stabilization (DNS).

The main question it aims to answer is:

* Which of these three exercises produces the highest activity in the quadriceps muscles (Vastus medialis, Vastus lateralis, and Rectus femoris)?
* Researchers will compare all three exercises to see which one best activates the quadriceps muscles.

Participants will:

* Perform all three exercises in a random order
* Have sensors (surface EMG) placed on the Vastus medialis, Vastus lateralis, and Rectus femoris muscles to record activity
* Complete each exercise with standardized timing

This information may help guide training and injury prevention programs for fencing athletes by identifying which exercises most effectively activate the quadriceps muscles.

DETAILED DESCRIPTION:
This study aims to compare the effects of three exercises-single-leg decline squat, single-leg decline squat with core activation, and Dynamic Neuromuscular Stabilization (DNS)-based half high kneeling exercise-on quadriceps muscle activity in fencers. Fencing involves asymmetric movements that demand high neuromuscular coordination, strength, and power, particularly in the lower extremities. The lunge, a key movement, relies on horizontal peak velocity influenced by back leg extensor strength and power. Lumbopelvic stability is crucial for injury prevention and performance enhancement, as it stabilizes the body against external stresses and optimizes joint function.DNS, grounded in neurodevelopmental kinesiology, focuses on activating the integrated spinal stabilization system (ISSS), which includes intersegmental spinal muscles, deep neck flexors, diaphragm, abdominal wall, and pelvic floor muscles. This approach integrates optimal breathing patterns, improves movement quality, and ensures functional joint centration to maximize strength efficiency and minimize mechanical stress.The protocol involves electromyographic (EMG) assessment of the vastus medialis obliquus (VMO), vastus lateralis (VL), and rectus femoris (RF) muscles on the dominant side during the exercises. Participants, aged 18-24 years with at least 5 years of fencing experience and no recent knee injuries or DNS training, undergo assessments in a controlled laboratory setting.Surface EMG is recorded using an eight-channel system (Noraxon, USA) with a sampling frequency of 1500 Hz. Electrode placement follows SENIAM recommendations: VMO at 80% of the distance between the anterior border of the medial collateral ligament and the superior anterior iliac spine; VL at two-thirds along the line from the anterior superior iliac spine to the lateral patella edge; RF at the midpoint between the anterior superior iliac spine and the upper patella edge. Skin preparation ensures impedance below 2 kΩ. Maximum voluntary isometric contraction (MVIC) testing normalizes EMG data, performed seated with hips at 90° and knees at 60° flexion, involving three 5-second maximal contractions with 30-second rests.Exercises are randomized and performed with a metronome at 60 beats per minute to standardize 3-second concentric, isometric, and eccentric phases per repetition. Three trials per exercise are conducted, with 30-second rests between trials. Single-leg decline squat: Performed on a 25° decline board, dominant leg only, to 60° knee flexion, with an adjustable mechanical device for depth control.

Single-leg decline squat with core activation: Identical to the above, plus abdominal bracing to enhance trunk stability, mimicking ISSS activation.

DNS-based half high kneeling: Involves forward leg at 90° hip/knee flexion with slight abduction/external rotation, contralateral knee on ground; posterior shift maintains ISSS activation, neutral pelvis, and spinal alignment, with tactile cues from the investigator.

All EMG data will be stored for offline processing. Raw EMG signals will be filtered using appropriate band-pass filters to remove movement artifacts and high-frequency noise. The filtered EMG signals will then be rectified and smoothed (for example, by calculating the root mean square over a defined moving window). For each participant, normalized EMG amplitude (%MVIC) for each muscle and each exercise will be calculated by averaging across the repetitions and across the predefined movement cycle. These normalized values for vastus medialis, vastus lateralis, and rectus femoris will form the basis of the primary analyses comparing the three exercises.

Planned statistical analyses will use within-subject methods appropriate for repeated measures (for example, repeated-measures ANOVA or non-parametric equivalents, depending on data distribution). Assumptions of the selected statistical tests (such as normality) will be checked, and corrections will be applied as needed. The comparisons of interest will focus on differences in normalized quadriceps muscle activity between the three exercises for each of the recorded muscles. Effect sizes and confidence intervals may be calculated to describe the magnitude and precision of differences. No interim analyses or long-term follow-up are planned, as this is a single-session study.

ELIGIBILITY:
Inclusion Criteria:

* Practicing fencing for at least 5 years
* Age between 18 and 24 years
* No systemic or neurological problems
* No knee pain on the dominant side

Exclusion Criteria:

* History of knee injury in the past year
* History of surgery on the dominant lower extremity
* History of patellar tendinitis
* Previous experience with Dynamic Neuromuscular Stabilization (DNS) training
* Pain while performing exercises during the test protocol

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Normalized quadriceps muscle activation measured by surface electromyography (EMG) | Through study completion, an average of 1 year".
  Quadriceps muscle activation will be assessed in the dominant leg using surface electromyography (EMG) during three different exercises (single-leg decline squat, single-leg decline squat with core activation, and DNS-based half high-kneeling exercise). Bipolar surface EMG electrodes will be placed over the vastus medialis, vastus lateralis, and rectus femoris muscles according to standard recommendations.
  Raw EMG signals will be filtered, rectified, and converted to root mean square (RMS) values. For each muscle and each exercise, EMG amplitudes will be normalized to the corresponding maximal voluntary isometric contraction (MVIC) and expressed as a percentage of MVIC (%MVIC). The primary outcome will be the average normalized EMG amplitude (%MVIC) recorded during the repetitions of each exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Bicici Ulusahin, PT PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Gazi University Health Sciences Faculty, Sports Rehabilitation Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
(%MVIC for vastus medialis obliquus, vastus lateralis, and rectus femoris during each exercise condition and contraction phase), will be shared.
  Data will be shared upon reasonable request to the corresponding author. Requests must include a methodologically sound proposal, and a data use agreement will be required.
Supporting Information: Study Protocol, SAP
Time Frame: Available 6 months after publication of the main results.
Access Criteria: Documents will be shared upon reasonable request to the corresponding author.
URL: https://clinicaltrials.gov/NotAvailable